CLINICAL TRIAL: NCT04088851
Title: "Non-invasive Measurement of Hepatic Substrate Flux Rates in People with Diabetes Mellitus Type 2"
Brief Title: "Hepatic Substrate Flux Rates in Type 2 Diabetes"
Acronym: IMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IMPACT
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes, redox shuttle, gluconeogenesis
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin - T2D (Experimental): Participants with type-2 diabetes will intake metformin 1 g daily for 2 weeks
  Interventions: Drug: On Metformin
- No Metformin - T2D (Placebo Comparator): Participants with type-2 diabetes will pause metformin 1 g daily for 2 weeks
  Interventions: Drug: Off Metformin

INTERVENTIONS:
Drug: On Metformin — Oral intake of Metformin (1 g / day) for 2 weeks
  Arms: Metformin - T2D
Drug: Off Metformin — No oral intake of Metformin (1 g / day) for 2 weeks
  Arms: No Metformin - T2D

SUMMARY:
Investigation of the effects of redox shuttle inhibition by metformin on gluconeogenic flux rates of lactate and glycerol in humans with type 2 diabetes

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is characterized by insulin resistance and relative insulin deficiency leading to hyperglycemia. Enhanced endogenous glucose production during fasting is a key feature of hepatic insulin resistance and a major contributor to deterioration of glycemia. Metformin reduces fasting gluconeogenesis (GNG); the underlying mechanisms are still not fully understood, but involve the inhibition of complexes of the electron transport chain and thus the redox shuttle.

The investigators have previously provided evidence for abnormal hepatic ATP synthesis and mitochondrial efficiency in T2D, but it remains unknown, how and which substrate fluxes account for excessive GNG in T2D. For this reason, this proposal aims at investigating hepatic glucose and energy fluxes in T2D with focus on gluconeogenic contribution of lactate and glycerol to hepatic mitochondrial substrate flux, mitochondrial ATP synthase flux and the activity of the redox shuttle, also after metformin intake, by using a novel combination of positional isotopomer nuclear magnetic resonance (NMR) analysis (PINTA) with multinuclei magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion criteria:

* type 2 diabetes (duration <7 years),
* age (18-75 years)
* BMI <40 kg/m2
* HbA1c 6-15%

Exclusion criteria:

* uncontrolled hyperglycaemia (>340 mg/dl)
* diabetes types other than type 2 diabetes (ADA criteria)
* thiazolidinedione use during the preceding 6 months
* clinically relevant angiopathy, restrictive or obstructive lung diseases
* other acute or chronic diseases including wounds and the use of pharmacological agents known to affect insulin sensitivity, lipid metabolism or immunological function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic gluconeogenic flux (U-13C-lactate tracer) (mg/min) | 2 weeks
  Hepatic gluconeogenic flux rates from lactate [mg/min] in humans with T2D w/wo metformin treatment will be measured by specific tracer metabolism and turnover of the substrates.
Hepatic gluconeogenic flux (glycerol tracer) (mg/min) | 2 weeks
  Hepatic gluconeogenic flux rates from glycerol [mg/min] in humans with T2D w/wo metformin treatment will be measured by specific tracer metabolism and turnover of the substrates.

SECONDARY OUTCOMES:
Endogenous glucose production (mg/min/kg BW) | 2 weeks
  Endogenous glucose production (mg/min/kg BW) in humans with T2D w/wo metformin treatment will be measured by specific tracer metabolism and turnover of the substrates.
Hepatic mitochondrial oxidative flux (mg/min) | 2 weeks
  Hepatic mitochondrial oxidative flux (mg/min) in humans with T2D w/wo metformin treatment will be measured by specific tracer metabolism and turnover of the substrates.
Hepatic gammaATP (mmol/L) | 2 weeks
  Hepatic energy [ATP mmol/l] content will be assessed in people with T2D with and without metformin treatment by employing specific 31P- magnetic resonance spectroscopy.
Hepatic lipid content (%) | 2 weeks
  Hepatic fat [%] content will be assessed in people with T2D with and without metformin treatment by employing specific 1H- magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No